CLINICAL TRIAL: NCT04602624
Title: An Open-Label Evaluation of the Safety and Tolerability of SAGE-718 in Participants With Mild Cognitive Impairment or Mild Dementia Due to Alzheimer's Disease
Brief Title: A Study to Evaluate the Safety and Tolerability of SAGE-718 in Participants With Mild Cognitive Impairment or Mild Dementia Due to Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 718-CNA-201
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease; Cognitive Dysfunction; Mild Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAGE-718 (Experimental): Participants received SAGE-718 3 mg oral tablets, once daily in the morning for 14 days.
  Interventions: Drug: SAGE-718

INTERVENTIONS:
Drug: SAGE-718 — SAGE-718 oral tablets.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of SAGE-718 and its effects on cognitive and neuropsychiatric symptoms in participants with mild cognitive impairment (MCI) or mild dementia due to Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Participant meets the following criteria for MCI or mild dementia due to AD at Screening: has a memory complaint, has clinical dementia rating (CDR) score of 0.5 to 1.0 (inclusive) with a memory box score ≥0.5, has essentially preserved activities of daily living
2. Participant has a score of 15 to 24 (inclusive) on the Montreal Cognitive Assessment at Screening
3. Participant has normal premorbid intelligence quotient (IQ) at Screening
4. Participant has a study partner who is reliable, competent, at least 18 years of age, willing to be available to the study center by phone, support study-specific activities, and accompany the participant to study visits as needed

Exclusion Criteria:

1. Participant has any medical or neurological condition (other than AD) that might be contributing to the participant's cognitive impairment or history of cognitive decline
2. Participant has a history of brain surgery, deep brain stimulation, a significant head injury causing loss of consciousness greater than 30 minutes, or hospitalization due to a brain injury
3. Participant has a history, presence, and/or current evidence of a clinically-significant intracranial abnormality (eg, stroke, hemorrhage, space-occupying lesion) that could account for the observed cognitive impairment (excluding abnormalities consistent with underlying AD pathology)
4. Participant has a history of possible or probable cerebral amyloid angiopathy, according to the Boston Criteria
5. Participant has a history of seizures or epilepsy, with the exception of a single episode of febrile seizures in childhood
6. Participant has current or recent suicidality

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Sage Investigational Site, Phoenix, Arizona
  - Sage Investigational Site, Redlands, California
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, St. Petersburg, Florida
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Gaithersburg, Maryland
  - Sage Investigational Site, Farmington Hills, Michigan
  - Sage Investigational Site, Omaha, Nebraska
  - Sage Investigational Site, North Canton, Ohio

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at investigative sites in the United States from 07 December 2020 to 28 September 2021.
Pre-assignment Details: A total of 58 participants were screened, of which 26 participants were enrolled to receive SAGE-718.
Period: Overall Study
Arm/Group | SAGE-718
Started | 26
Completed | 24
Not Completed | 2
Not completed — Protocol Deviation | 1
Not completed — Withdrawal by Participant | 1

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were administered investigational product (IP).
Arm/Group | SAGE-718
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 4
  Race: White | 21
  Race: Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered with a pharmaceutical product and that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an IP whether or not related to the product. An AE can include any undesirable medical condition, even if no study treatment has been administered. TEAEs were defined as an AE with an onset date on or after the date of the first dose of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: From first dose of study drug up to last follow up visit (up to 28 days)
Population: Safety Set included all participants who were administered IP.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-718
Number analyzed (Participants) | 26
Participants | 7

2. Secondary Outcome: Percentage of Participants With at Least One Potentially Clinically Significant (PCS) Change in Vital Signs Measurements
Description: PCS changes for vital signs included: Supine Systolic Blood Pressure (SBP) >180 millimeters of mercury (mmHg), SBP decrease from baseline of ≥ 30 mmHg, standing 1-minute SBP >180 mmHg, standing 3 minutes SBP decrease from baseline of ≥ 30 mmHg, Supine diastolic BP (DBP) decrease from baseline of ≥ 20 mmHg, standing 1-minute DBP decrease from baseline of ≥ 20 mmHg, standing 1-minute DBP increase from baseline of ≥ 20 mmHg, standing 3-minute DBP increase from baseline of ≥ 20 mmHg, orthostatic SBP: supine-1 minute standing ≥ 20 mmHg and supine-3 minute standing ≥ 20 mmHg, orthostatic DBP: supine-1 minute standing ≥ 10 mmHg and supine-3 minute standing ≥ 10 mmHg. Percentage of participants with at least one PCS change in vital signs measurements were reported.
Time Frame: From first dose of study drug up to last follow-up visit (up to 28 days)
Population: Safety Set included all participants who were administered IP. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Number; unit: percentage of participants
Arm/Group | SAGE-718
Number analyzed (Participants) | 25
percentage of participants | 64.0

3. Secondary Outcome: Percentage of Participants With at Least One Potentially Clinically Significant Change in Laboratory Assessments
Description: PCS changes for laboratory assessments included: hematology: hematocrit- male low (<0.385 fractions of 1), hemoglobin male low (<115 grams per liter [g/L]) and biochemistry: glucose high (>13.9 millimoles per liter [mmol/L]), potassium low (<3.3 mmol/L), blood urea nitrogen high (>10.71 mmol/L)., Percentage of participants with at least one PCS change in laboratory assessments were reported.
Time Frame: From first dose of study drug up to last follow-up visit (up to 28 days)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | SAGE-718
Number analyzed (Participants) | 25
percentage of participants
  Hematology | 12.0
  Biochemistry | 16.0

4. Secondary Outcome: Percentage of Participants With at Least One Potentially Clinically Significant Change in Electrocardiogram (ECG) Measurements
Description: PCS changes for ECG measurements included: QTcF Interval >450 to ≤480 milliseconds (msec), >480 to ≤500 msec, and ≥30 to ≤60 msec increase from baseline. Percentage of participants with at least one PCS change in ECG measurements were reported.
Time Frame: From first dose of study drug up to last follow-up visit (up to 28 days)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | SAGE-718
Number analyzed (Participants) | 25
percentage of participants | 32.0

5. Secondary Outcome: Percentage of Participants With Suicidal Ideation or Behavior Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS scale assesses the lifetime experience of participants with suicidal ideation (SI) and suicidal behavior (SB). The C-SSRS included "yes" or "no" responses for assessment of suicidal ideation and behavior as well as numeric ratings for the severity of ideation, if present (with score range from 1 to 5, with 5 being the most severe). The C-SSRS SI items involved wish to be dead, non-specific active suicidal thoughts, active SI with any methods, active SI with some intent and active SI with a specific plan. The C-SSRS SB items involved preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt (non-fatal) and completed suicide. Percentage of participants with a response of 'yes' for suicidal ideation or behavior were reported.
Time Frame: Up to Day 28
Population: Safety Set included all participants who were administered IP.
Measure: Number; unit: percentage of participants
Arm/Group | SAGE-718
Number analyzed (Participants) | 26
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Screening up to last follow-up visit (approximately 49 days)
Description: Safety Set included all participants who were administered IP.
Arm/Group | SAGE-718
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 7/26
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAGE-718 (N=26)
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT04602624/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04602624/SAP_001.pdf